CLINICAL TRIAL: NCT05588492
Title: The Safety, Completion Rate and Prevention Effect by Rifamycin-containing Regimens for Latent Tuberculosis Infection in Patients With Kidney Transplantation: a Prospective Intervention Pilot Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 202110073MIND
Record Dates: First submitted 2022-05-03; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-04

CONDITIONS: Pulmonology
Keywords: latent tuberculosis infection,mycobacterium tuberculosis
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifamycin containing regimen (Experimental): Rifamycin containing regimen
  Interventions: Drug: Rifamycin-containing regimen
- Rifamycin-free regimen (Experimental): Rifamycin-free regimen
  Interventions: Drug: Rifamycin-free regimen

INTERVENTIONS:
Drug: Rifamycin-containing regimen — Rifamycin-containing regimen
  Arms: Rifamycin containing regimen
Drug: Rifamycin-free regimen — Rifamycin-free regimen
  Arms: Rifamycin-free regimen

SUMMARY:
Tuberculosis (TB) remains the leading infectious disease worldwide and kidney transplant recipients (KTR) is high risk population needing prevention from reactivation, which cause high mortality. In fact, its latent tuberculosis infection (LTBI) is increasing after transplantation and has been identified as a risk factor for TB. However, the suitable regimen for LTBI treatment in KTRs remains unclear. Currently, three-month rifamycin-containing regimens, such as weekly rifapentine and isoniazid (3HP) or daily rifampicin and isoniazid (3HP), are common because its non-inferiority to nine-month of daily isoniazid (9H) and high completion rate by its short course in TB contacts. However, KTRs have many differences from general population, like use of immune-suppressants and possible residual renal insufficiency, so that to prescribe rifamycin-containing LTBI treatment regimens may have many concerns. One biggest concern is that drug-drug interaction between rifamycin and immunosuppressants. In addition, there is no study before in investigating the use of rifamycin-containing regimen in the population of KTRs (only study for kidney transplant candidates).

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the leading infectious disease worldwide and kidney transplant recipients (KTR) is high risk population needing prevention from reactivation, which cause high mortality. In fact, its latent tuberculosis infection (LTBI) is increasing after transplantation and has been identified as a risk factor for TB. However, the suitable regimen for LTBI treatment in KTRs remains unclear. Currently, three-month rifamycin-containing regimens, such as weekly rifapentine and isoniazid (3HP) or daily rifampicin and isoniazid (3HP), are common because its non-inferiority to nine-month of daily isoniazid (9H) and high completion rate by its short course in TB contacts. However, KTRs have many differences from general population, like use of immune-suppressants and possible residual renal insufficiency, so that to prescribe rifamycin-containing LTBI treatment regimens may have many concerns. One biggest concern is that drug-drug interaction between rifamycin and immunosuppressants. In addition, there is no study before in investigating the use of rifamycin-containing regimen in the population of KTRs (only study for kidney transplant candidates). Therefore, we conducted this project aiming to monitor the safe issues (adverse events and drug-drug interaction), completion rate, and prevention effect in the population of KTRs.

ELIGIBILITY:
Inclusion Criteria:

1. Received kidney transplant, and
2. Will receive interferon-gamma release assay (IGRA) for LTBI, and
3. If IGRA was positive, participants agree to receive LTBI treatment

Exclusion Criteria:

1. Age < 20 years old
2. pregnancy
3. Suspicious active tuberculosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | up to 12 months
  Incidence of treatment related any adverse event

SECONDARY OUTCOMES:
Secondary Outcome Measure | up to 12 months
  proportion of treatment interruption

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan